CLINICAL TRIAL: NCT02404363
Title: A Phase III Multi-centre Double-blind Placebo Controlled Study Analysing the Efficacy and Safety of Daily Administration of a P2Y12 Inhibitor (Clopidogrel) for the Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Safety and Efficacy of Clopidogrel in Locally Advanced and Metastatic Pancreatic Adenocarcinoma Treated With Chemotherapy
Acronym: PANCREADOGREL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment problem
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Francophone Thrombose et Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P130936; 2014-001463-12 (EudraCT Number)
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Locally Advanced Pancreatic Cancer; Adenocarcinoma, Pancreas; Metastatic Pancreatic Cancer
Keywords: Clopidogrel; Pancreatic Cancer; Efficacy; Chemotherapy; Microparticles; Disease free survival; First line chemotherapy
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Clopidogrel tablets 75 mg for six months:
  Interventions: Drug: Clopidogrel
- Comparator (Placebo Comparator): Placebo tablet 75 mg for six months:
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel tablets 75 mg for six months:
  In case of treatment with aspirin < or = 75 mg/d or prophylactic LMWH --> clopidogrel 75 mg/d If aspirin = 0 + LMWH = 0 --> clopidogrel 150 mg/d x 7days then 75mg/d
  Arms: Clopidogrel
Drug: Placebo — Placebo tablets 75 mg for six months:
  In case of treatment with aspirin < or = 75 mg/d or prophylactic LMWH --> placebo 75 mg/d If aspirin = 0 + LMWH = 0 --> placebo 150 mg/d x 7days then 75mg/d
  Arms: Comparator

SUMMARY:
Clopidogrel has been shown to slow down tumor progression in orthoptic pancreatic murine tumor.

In a pilot study, the rate of microparticles was correlated with response rate of pancreatic adenocarcinoma.

The aim of the study is;

* to compare the phenotypes of coagulation, the tumor progression and metastasis formation with and without clopidogrel treatment in association with chemotherapy in advanced pancreatic cancer patients
* to correlate the decrease of microparticles levels after one month of chemotherapy with tumor response (ancillary study)

DETAILED DESCRIPTION:
Several studies have been performed to understand the cellular mechanisms involved in the development of VTE in cancer patients. The pathogenesis of a thrombotic state is linked to the presence of a tumor and is associated with the development of a hypercoagulant state, namely coagulopathy, which confers numerous advantages to the cancer cells. Indeed, both activation of the coagulation cascade and aggregation of blood platelets around cancer cells protect themselves from the immune response; facilitate their circulation in the bloodstream and their adhesion at potential sites of metastasis. Beside its implication in the activation of coagulation, the TF/FVIIa complex also influences pathways that activate cell-bound protease activated receptors (PARs) leading to the activation of inflammatory and angiogenic responses. Furthermore, a soluble variant of TF, known as alternatively spliced TF (asTF) stimulates angiogenesis independent of FVIIa. This leads to a model in which the presence of Tissue Factor (TF), generation of thrombin and platelets activation all directly participate to the cancer progression and dissemination. The presence of TF and the activation of platelets participate to the progression of the tumor.

A retrospective study collected clinical information and plasma samples of 117 patients with pancreatic or biliary cancer, of which 68% were pancreatic cancer and 29% biliary cancers. Thrombotic events occurred in 52 (44.4%) patients. Mean and median tissue factor for all patients were 2.15 pg/mL and 1.20 pg/mL, respectively (range: 0.17-31.01 pg/mL). Elevated Tissue Factor levels were significantly associated with VTE events (P=0.04), and an elevated tissue Factor level was associated with a worse overall survival (hazard ratio, HR: 1.05; P=0.01).

This procoagulant state could be due to the expression of active TF and transmembrane proteins (PSGL-1, Muc1, …) by the cancer cell itself or cancer cell-derived microparticles leading to platelets activation and aggregation. While studying the key role of TF bearing cancer cell-derived microparticles in cancer associated thrombosis, the investigators have previously shown (Dubois C, INSERM UMR 1076 Marseille) that both endogenously generated and exogenously injected pancreatic cancer cell-derived microparticles expressing TF (PancO2), but not their parental tumor cells, accumulated at the site of injury in a P-selectin dependent manner. Their presence directly correlates with the size of the thrombus. Based on these data, the investigators first hypothesized that treatment with anticoagulant and / or antiplatelet drugs may prevent tumor progression and formation of metastasis, as well as thrombosis associated cancer, in addition to prevention of coagulopathy.

Then Dubois & al compared the effect of an inhibitor of platelet activation, Clopidogrel, and an inhibitor of the activation of the coagulant cascade, low molecular weight heparin (LMWH) on tumor growth and thrombosis associated with cancer. Concentrations of drugs used were calculated to induce a 50% reduction of thrombus formation following a laser-induced injury in healthy mice. A diminution of kinetics of tumor growth was observed in mice treated by the 2 drugs in comparison with non-treated mice. Twenty days following injection of cancer cells, the volume of the tumor was reduced by 85% and 87% when LMHW or Clopidogrel were used, respectively. However, kinetics of tumor growth and volumes of tumors 20 days post-injection were similar in mice treated by Clopidogrel in presence or absence of pathological TF expressed by cancer cells.

Cancer cell-derived microparticles are responsible for the thrombotic phenotype observed in mice developing a cancer via interactions between P-selectin expressed by aggregating platelets and activated endothelium and PSGL-1 present at the surface of cancer cell-derived microparticles. Before injury but after their infusion in bloodstream, exogenous labeled cancer cell-derived microparticles were detected in the cremaster microcirculation of non-treated or Clopidogrel treated mice. However, following an injury, cancer cell-derived microparticles were accumulating at the site of thrombus formation only in non-treated mice bearing a PancO2-LowTF or High TF tumor. Tissue Factor (TF) is both a main effector of the coagulation cascade and a protein involved in the development of solid tumors. In vivo, following a laser-induced injury, the activation of the endothelial wall, as well as the presence of activated platelets, are the main source of P-selectin. The quantity of P-selectin present at the site of injury was 4 fold less important in mice bearing a PancO2 tumor and treated by Clopidogrel in comparison with non-treated mice. Interestingly, PanCO2 cancer cell-derived microparticles express both TF and TFPI (Tissue Factor Inhibitor), a biological inhibitor of the coagulation cascade in an active form. To confirm that cancer-cell derived microparticles may participate in the inhibition of the blood coagulation observed when the pathological TF is shut down, the investigators compared fibrin generation at the site of injury in PancO2-High TF and Low-TF cancer mice in presence of absence of Clopidogrel.

Fibrin formation at the site of laser-induced injury was significantly more important (P<0,01) in mice following injection of Panc02-High TF in comparison with wild type mice. Treatment of these mice by Clopidogrel diminished the production of fibrin at a level comparable to the ones observed in wild type mice. When the pathological TF was shut down, production of fibrin was strongly reduced in comparison with both the group of mice injected by Panc02 cells and the group of wild type mice. the investigators conclude that when cancer cells and cancer cell-derived microparticles express active TF, their incorporation to a growing thrombus participates to the generation of a thrombotic phenotype. When TF expressed by cancer cells is shut down, cancer cells microparticles still incorporate at the site of thrombus formation, but reduces activation of TF, inhibiting fibrin generation and thrombus formation by bringing TFPI at the site of injury.

Based on observations, the investigators hypothesized that inhibition of platelet activation by reducing both thrombosis associated with cancer and tumor growth could constitute an interesting therapy to treated cancer and thrombosis. To test the hypothesis the investigators then developed a syngeneic orthoptic model of pancreatic cancer and could confirm that when mice were treated with Clopidogrel or Aspirin, the growth of the primary tumor was significantly reduced and the development of metastasis was limited (Mege et al.). However the benefit from aspirin was observed in mice only when treated immediately at time of onset of cancer, id est when injection of cancer cells were performed. On the contrary, the effects of clopidogrel were obtained independently of the tumor size, and tumor development or onset and even once cancer was at an advanced stage. Altogether with the action of anti-platelet drugs on thrombosis, these results indicate that Clopidogrel does represent a promising therapeutic drug to limit thrombosis and reduce the development of tumors and metastasis.

The investigators showed in the experimental model that TF expressed by cancer cells was involved in thrombosis associated with a cancer and in the growth of the tumor in vivo. Beside its functions in coagulation, TF was also described following phosphorylation and binding of its cytoplasmic tail to filamin, to induce transcriptional activation of different growth factors, including VEGF. This intracellular pathway may also participate in the growth of the tumor, but also in angiogenesis. Furthermore, TF expression was also reported to influence motility, survival and proliferation of cancer cells via the activation of PAR-1 and PAR-2, although in this study proliferation of Panc02 cells were not affected by inhibition of TF expression. Cancer cells may directly activate platelets by secreting ADP, Thromboxane A2 and MMP-2 (Matrix Metallo Proteinase 2) and express at their surface ligands to platelets, such as PSGL-1. In bloodstream, this leads to an aggregation of platelets around cancer cells described to protect them from destruction by the immune system, blood shear stress and to facilitate cancer cells interactions with the endothelium. However, the direct involvement of these platelet agonists was not demonstrated in vivo. When mice were treated with LMWH, a decrease in tumor development was observed similar to the ones obtained when pathological TF was shut down. Also, treatment by Clopidogrel did not significantly affect the growth of the tumor in the group of Panc02 miRNA TF mice or in the group of Panc02 mice treated by LMWH. This strongly suggests that activation of platelets is involved in the growth of the tumor, but also that the main activator of platelet is TF expressed by cancer cells and nor ADP nor Thromboxane A2. These secondary agonists may be involved when secreted as a consequence of platelet activation generated by thrombin through a TF dependent pathway. Last, they may play an important role not directly in the growth of the tumor, but rather in the formation of metastasis when cancer cells have to be present in the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Locally advanced or metastatic pancreatic cancer
* Measurable primary pancreatic cancer or metastasis
* No previous chemotherapy either in an adjuvant or metastatic setting
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate bone marrow: granulocyte count ≥ 1.5 G/L; and platelet count ≥ 100 G/L
* Adequate liver function: bilirubin ≤ 2 times the upper limit of the normal range, transaminases (AST and ALT) ≤ 3 times the upper limit of the normal range
* Adequate renal function: calculated clearance rate > 60 m.mn-1 (Estimated glomerular filtration rate using Modification of Diet in Renal Disease (MDRD) formula or Cockcroft-Gault formula)
* Women of childbearing potential must use an effective birth control method

Exclusion Criteria:

* Endocrine or acinar pancreatic carcinoma
* Pancreatic metastasis of other primary tumors
* Previous radiotherapy for measurable lesions
* Previous chemotherapy
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis
* Other prior malignancy. Adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or any other cancer from which the patient has been disease free for > 5 years are allowed.
* Known HIV disease requiring antiretroviral treatment
* Hemorrhagic diathesis
* Aspirin with a daily dose > 75 mg
* Curative dose of LMWH
* Recent venous thromboembolism (< 1 year)
* Patients under VKA
* Lesion of the digestive tract that could be hemorrhagic with clopidogrel treatment
* Active infection
* Chronic diarrhea
* Cardiac disease with a left ventricular ejection fraction below 45%
* Hypersensitivity to clopidogrel or its excipients
* Patients with severe hepatic impairment
* Patients who are pregnant or breast feeding, or who are not using effective birth control methods
* Participation in another clinical research protocol, participation in a trial of routine care is authorized at the same time as PANCREADOGREL
* Patient under tutorship or curatorship
* Patients unwilling or unable to comply with the protocol
* Not affiliated to health system ("bénéficiaire ou ayant droit")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Response to treatment based on RECIST 1.1 criterion | up to 6 months
  Progression free survival

SECONDARY OUTCOMES:
Venous thromboembolic events | up to 12 months
  Diagnosis of pulmonary embolism (PE), deep venous thrombosis (DVT) and visceral vein event.
Response to treatment based on RECIST 1.1 criterion | up to 12 months
  Overall response rate
Overall survival | up to 12 months
  Overall survival is defined as time from randomization to death from any cause
Bleedings | up to 12 months
  All suspected bleedings will be classified as major, minor, clinically relevant non-major or no bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DEBOURDEAU, MD, Principal Investigator — Institut Sainte Catherine - Avignon
Locations (1):
- Service d'oncologie digestive - Institut Sainte Catherine, Avignon, France